CLINICAL TRIAL: NCT07204067
Title: Effectiveness of Mirror Therapy in Improving Motor Recovery and Hand Function in Patients With Acute Stroke A Randomized Controlled Trial
Brief Title: Mirror Therapy for Hand Function Recovery in Acute Stroke
Acronym: Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RIPHAH-REC Sapna Kursheed
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Stroke
Keywords: Mirror Therapy Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Parallel Assignment (2 arms)
Who Masked: Participant
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy + Conventional Physiotherapy (Experimental): Experimental: Mirror Therapy + Conventional Physiotherapy
  Device/Procedure: Mirror Therapy (20 min/session) + immediate Conventional Physiotherapy (20 min/session)
  Schedule: 2 sessions/week for 1 week (total: 2 sessions)
  MT Procedure: Mirror (box or plain) placed along mid-sagittal plane reflecting the non-paretic limb while hiding the paretic limb. Participants perform bilateral symmetrical movements focusing on the mirror image (e.g., wrist flex/ext, finger flex/ext, elbow flex/ext, reaching & grasping).
  Conventional Content (immediately after MT): strengthening & functional task practice (e.g., reaching/transfers), plus targeted hand training: theraputty squeezes, finger extension with rubber band, towel wringing, lifting small objects, reaching overhead/side-to-side with weight, weighted ball toss/catch.
  Interventions: Behavioral: Mirror Therapy Conventional Physiotherapy
- Conventional Physiotherapy Only (Active Comparator): Procedure: Conventional Physiotherapy (20 min/session), no mirror. Same schedule and exercise menu as above without visual mirror feedback.
  Notes: The proposal specifies 1 week duration with 2 sessions/week, 20 min each; centers may extend to clinically standard dosage via protocol amendment if needed.
  Interventions: Behavioral: Mirror Therapy Conventional Physiotherapy

INTERVENTIONS:
Behavioral: Mirror Therapy Conventional Physiotherapy — Experimental: Mirror Therapy + Conventional Physiotherapy Mirror therapy performed 20 min/session, 2 sessions/week for 1 week. A mirror is placed midsagittal, reflecting the non-paretic limb while hiding the paretic limb. Patients perform bilateral movements (wrist, finger, elbow flex/extension; reaching/grasping) while focusing on the mirror image. This is followed by 20 min of conventional physiotherapy, including strengthening, functional tasks, theraputty squeezes, finger extension with rubber band, towel wringing, lifting small objects, overhead reaching, and ball toss.
  Active Comparator: Conventional Physiotherapy Only Conventional physiotherapy 20 min/session, 2 sessions/week for 1 week. Exercises include upper limb strengthening, functional task practice, theraputty squeezes, finger extension with rubber band, towel wringing, lifting small objects, overhead reaching, and ball toss.
  Other Names: intervention for stroke

SUMMARY:
Randomized controlled trial to determine whether mirror therapy (MT), added to conventional physiotherapy, improves upper-limb motor recovery, hand function, spasticity, and range of motion (ROM) in acute stroke compared with conventional physiotherapy alone. Outcomes include ARAT, Motor Assessment Scale, Modified Ashworth Scale, and goniometric ROM.

DETAILED DESCRIPTION:
Stroke causes significant upper-limb impairment in the acute stage; early, targeted rehabilitation leverages heightened neuroplasticity. Mirror therapy uses a mid-sagittal mirror to reflect movements of the non-paretic limb, creating the illusion of normal movement in the paretic limb, recruiting mirror neuron circuits and facilitating motor relearning. Prior work suggests MT can improve fine and gross motor skills, reduce spasticity, and increase active ROM. This trial operationalizes a pragmatic MT protocol integrated with standard inpatient/outpatient physiotherapy in acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-55 years
* Acute ischemic or hemorrhagic stroke within the last 1 month
* Unilateral hemiparesis/hemiplegia
* Medically stable and cleared for rehabilitation
* Able to follow verbal instructions; MMSE ≥ 24
* Provides written informed consent

Exclusion Criteria:

* Recurrent stroke or bilateral involvement
* Severe cognitive impairment (MMSE < 24)
* Visual field deficits, unilateral neglect, or severe aphasia interfering with MT
* Other neurological disorders (e.g., Parkinson's, MS)
* Orthopedic conditions affecting upper limb/trunk
* Uncontrolled cardio-respiratory disease limiting exercise
* Severe spasticity (MAS ≥ 3) in affected limb
* Concurrent enrollment in other interventional trials
* Inability/refusal to consent

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-08-17 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Upper-Limb Function (ARAT total score, 0-57) | 6 Months
  Change from baseline to end of week 1; higher scores = better function.

SECONDARY OUTCOMES:
Motor Function (Motor Assessment Scale - relevant upper-limb items, 0-6 per item) | 6months
  Change baseline→week 1; higher = better.

OTHER OUTCOMES:
Spasticity (Modified Ashworth Scale, 0-4) | 6 months
  Change baseline→week 1; lower = less spasticity.
Range of Motion (Goniometric AROM at shoulder, elbow, wrist, finger joints; degrees) | 6 months
  Change baseline→week 1; higher = improved ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nadeem Ahmad, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University Malakand Campus, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No